CLINICAL TRIAL: NCT00880685
Title: Memantine Treatment of Kleptomania: An Open-Label Study
Brief Title: Memantine in the Treatment of Kleptomania
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0901M56882
Record Dates: First submitted 2009-03-18; First posted 2009-04-14 (Estimated); Results first posted 2014-03-05 (Estimated); Last update posted 2021-05-24 (Actual); Status verified 2021-04

CONDITIONS: Kleptomania
Keywords: Compulsive Stealing; Compulsive Shoplifting
MeSH Terms: conditions — Disruptive, Impulse Control, and Conduct Disorders | interventions — Memantine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Memantine (Experimental): Memantine 10-30mg
  Interventions: Drug: Memantine

INTERVENTIONS:
Drug: Memantine — 10-30mg, daily for 8 weeks
  Other Names: Namenda

SUMMARY:
The goal of the proposed study is to evaluate the efficacy and safety of memantine in kleptomania.

DETAILED DESCRIPTION:
The proposed study will consist of 8 weeks of treatment with memantine in 10 subjects with kleptomania. The hypothesis to be tested is that memantine will be effective in reducing the urges to steal in patients with kleptomania. The proposed study will provide needed data on the treatment of a disabling disorder that currently lacks a clearly effective treatment.

ELIGIBILITY:
Inclusion Criteria:

1. men and women age 18-65
2. current KM using the clinician-administered Structured Clinical Interview for Kleptomania (SCI-K)
3. stealing behavior within 2 weeks prior to enrollment.

Exclusion Criteria:

1. infrequent stealing (i.e. less than one time per week) that does not meet proposed criteria for kleptomania (KM)
2. unstable medical illness or clinically significant abnormalities on laboratory tests or physical examination at screen
3. history of seizures
4. myocardial infarction within 6 months
5. current pregnancy or lactation, or inadequate contraception in women of childbearing potential
6. a need for medication other than memantine with possible psychotropic effects or unfavorable interactions
7. clinically significant suicidality
8. current Axis I disorder determined by the Structured Clinical Interview for the DSM (SCID) and SCID-compatible modules for impulse control disorders (Grant et al., 2005), except for nicotine dependence
9. lifetime history of bipolar disorder type I or II, dementia, schizophrenia, or any psychotic disorder determined by SCID
10. current or recent (past 3 months) DSM-IV substance abuse or dependence
11. positive urine drug screen at screening
12. initiation of psychotherapy or behavior therapy within 3 months prior to study baseline
13. previous treatment with memantine; and 14) treatment with investigational medication or depot neuroleptics within 3 months, with fluoxetine within 6 weeks, or with other psychotropics within 2 weeks prior to study baseline.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-03; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon E Grant, MD, JD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Memantine 10mg-30mg: Memantine 10mg-30mg (active drug)
Period: Memantine 10mg
Arm/Group | Memantine 10mg-30mg
Started | 12
Completed | 10
Not Completed | 2
Not completed — Lost to Follow-up | 2
Period: Memantine 20mg
Arm/Group | Memantine 10mg-30mg
Started | 10
Completed | 9
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: Memantine 30mg
Arm/Group | Memantine 10mg-30mg
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Memantine 10mg-30mg
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.6 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Yale Brown Obsessive Compulsive Scale Modified for Kleptomania (KM-YBOCS)
Description: Scores could range from 0-40 with 0 being the least severe and 40 being the most severe. Here the total score was used. The Yale Brown Obsessive Compulsive Scale Modified for Kleptomania (KM-YBOCS) was completed at every visit (1-5), but the final visit (visit 5) will be the only score reported. The scale was given at baseline and weeks 2, 4, 6, and 8. Only the last visit (week 8) will be reported here.
Time Frame: Week 8 (last visit)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Memantine 10mg-30mg: Memantine 10mg-30mg (study drug)
Arm/Group | Memantine 10mg-30mg
Number analyzed (Participants) | 12
units on a scale | 5.4 (4.2)

2. Secondary Outcome: Kleptomania Symptom Assessment Scale (K-SAS)
Description: Scale used to measure severity of kleptomania. Scores could range from 0-36 with 0 being the least severe and 36 being the most severe. Here the total score was used. The K-SAS was completed at every visit (1-5), but the final visit (visit 5) will be the only score reported. The scale was given at baseline and weeks 2, 4, 6, and 8. Only the last visit (week 8) will be reported here.
Time Frame: Week 8 (last visit)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Memantine
Number analyzed (Participants) | 12
units on a scale | 12.3 (9.5)

3. Secondary Outcome: Clinical Global Impression Severity Scales (CGI)
Description: The overall impression of the clinician of the severity of the subject. Scores between 1 and 7 with 1 not being ill at all and 7 being one of the worst cases seen. CGI is given at baseline and weeks 2, 4, 6, and 8. Only the last visit (week 8) will be reported here.
Time Frame: Week 8 (last visit)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Memantine 10mg-30mg
Number analyzed (Participants) | 12
units on a scale | 2.2 (1.0)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the beginning of the study until study completion (3 years)
Groups:
- Memantine 10mg: Memantine 10mg (study drug)
- Memantine 20mg: Memantine 20mg (study drug)
- Memantine 30mg: Memantine 30mg (study drug)
Arm/Group | Memantine 10mg | Memantine 20mg | Memantine 30mg
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 3/12 | 4/10 | 2/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Memantine 10mg (N=12) | Memantine 20mg (N=10) | Memantine 30mg (N=9)
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Dry Mouth (General disorders) | 0 | 1 | 0
Increased Appetite (Metabolism and nutrition disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Dizziness (General disorders) | 1 | 1 | 1
Headache (Nervous system disorders) | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No